CLINICAL TRIAL: NCT06875167
Title: Semi-closed Loop Automated Insulin Therapy in the Pediatric Population Aged 2-6 Years With Type 1 Diabetes: Impact on Quality of Life and Glycemic Control
Acronym: Diablife
Status: Recruiting | Type: Observational
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Other Study IDs: 24-HPNCL-07 Diablife
Record Dates: First submitted 2025-03-04; First posted 2025-03-13 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Type 1 Diabetes; Closed Loop; Insulin; Quality of Life; Pediatric
Keywords: Closed-loop insulin therapy; type 1 Diabetic; Quality of life; pediatric patient
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study of the quality of life of diabetic children closed loop treatment versus other insulin therapy: Study of the quality of life of T1D children aged 2 to 6 years inclusive treated with a semi-closed loop insulin pump versus other types of insulin therapy. Each patient will be it's one controle.

SUMMARY:
The incidence of type 1 diabetes is increasing, with an incidence of +4% per year in France today.

The treatment for type 1 diabetes is insulin therapy. In recent years, new systems have emerged, so-called "semi-closed loop" systems, also called automated insulin therapy, which have proven their superiority in terms of quality of life and glycemic balance in adults and children over 6 years old.

Since January 24, 2024, the HAS now recognizes the indication of the semi-closed loop for the YPSOPUMP model in children aged 2 to 6 years. This is the first reimbursement in France of a closed loop system for the 2-6 year old age group. There are currently few studies comparing the quality of life of children in semi-closed loop versus other treatments (open loop or injections). Regarding quality of life, the studies found mainly concern the contribution for parents and the improvement of adolescents' sleep as in the study by Erin C Cobry et al from 2020 (6).

Our study therefore aims to demonstrate an improvement in quality of life but also in diabetes balance in type 1 diabetic patients on a closed loop insulin pump versus open loop or injections in the pediatric population aged 2-6 years.

ELIGIBILITY:
Inclusion Criteria:

* -Patients aged 2 to 6 years inclusive
* Presenting type 1 diabetes on insulin therapy
* Social security affiliates
* Patient initiating semi-closed loop treatment
* Family (at least one parent or representative of parental authority) agreeing to follow the training necessary for continuous measurement of glucose in real time.
* collection of non-opposition from one of the two parents or the representative of parental authority agreement

Exclusion Criteria:

* Opposition to participation in research involving humans or opposition to the use of data or samples and associated data (withdrawal of non-opposition).

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Type 1 Diabetic children aged 2 to 6 years treated with a semi-closed loop insulin pump at the Nice pediatric hospital
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
An improvement in the score on the general quality of life questionnaire in pediatrics PedsQL 4.0 which will be evaluated before the implementation of the semi-closed loop, at 1 month and 6 months after the implementation of the semi-closed loop. | the assessment of quality of life via the PedsQL 4.0 questionnaire will be evaluated before the implementation of the semi-closed loop, at 1 month and 6 months after the implementation of the semi-closed loop.
  The quality of life questionnaire includes 4 categories of questions regarding the last month: 1 category on physical capacity problems, 1 category on emotional state problems, 1 category on problems relating to others, and 1 category on problems with the community.
  Each category is rated from 0 (never) to 4 (almost always). The quality of life questionnaire intended for children aged 5 to 6 years concerns the last 7 days. The response is rated using a face scale (3 different faces) corresponding to the rating 0 (never), 2 (sometimes) and 4 (almost always).
  The overall quality of life of the diabetic child corresponds to the combined score of all the questions. The score range is 0 to 92, with lower scores indicating better quality of life.

SECONDARY OUTCOMES:
Compare the glycemic balance of patients on automated insulin therapy versus other treatments (open loop or injections) via TIR (time in range or time within the target). | The evaluation of the secondary criteria is carried out before the implementation of the semi-closed loop, then at 1 month and 6 months after implementation.
  Evolution of TIR (time in range or time in the target) when switching to semi-closed loop versus open loop.
Compare the glycemic balance of patients on automated insulin therapy versus other treatments (open loop or injections) via HbA1c. | The evaluation of the secondary criteria is carried out before the implementation of the semi-closed loop, then at 1 month and 6 months after implementation.
  Evolution of HbA1c during the transition to semi-closed loop versus open loop.
Compare the number of hypoglycemic episodes | The evaluation of the secondary criteria is carried out before the implementation of the semi-closed loop, then at 1 month and 6 months after implementation.
  Evolution of TUR (time spent in hypoglycemia) when switching to semi-closed loop versus open loop.
Compare time in hyperglycemia | The evaluation of the secondary criteria is carried out before the implementation of the semi-closed loop, then at 1 month and 6 months after implementation.
  Evolution of TAR (time spent in hyperglycemia) when switching to semi-closed loop versus open loop

CONTACTS AND LOCATIONS:
Overall Officials: Céline Gouillard-Darnaud, MD, Principal Investigator — Fondation Lenval
Locations (1):
- Fondation Lenval Hôpitaux pédiatrique Nice CHU Lenval, Nice, France, France

IPD SHARING:
Plan to Share IPD: Undecided